CLINICAL TRIAL: NCT02889679
Title: Underwater Resection of Non-pedunculated Colorectal Lesions: A Randomized Controlled Trial
Brief Title: Underwater Resection of Non-pedunculated Colorectal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Northern California Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-06-00766
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Neoplasms
Keywords: Colonoscopy; Polypectomy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Underwater resection (Experimental): All eligible lesion identified in a patient will be resected by the underwater technique. Excluded lesions will be resected by standard polypectomy.
  Interventions: Procedure: Underwater resection; Procedure: Standard polypectomy
- Conventional resection (Active Comparator): All eligible lesion identified in a patient will be resected by the conventional (gas distended colon) resection techniques. Excluded lesions will be resected by standard polypectomy.
  Interventions: Procedure: Conventional (gas distended colon) resection; Procedure: Standard polypectomy

INTERVENTIONS:
Procedure: Underwater resection — Underwater resection of eligible lesions will be performed with air exclusion (air will be suctioned and completely removed) without submucosal injection in a partially collapsed colon lumen filled with water. Water will be infused with the foot pedal to facilitate visualization during UR and there will be no limit to the amount of water infused. Hot and cold resection techniques will be utilized.
  Arms: Underwater resection
Procedure: Conventional (gas distended colon) resection — Conventional polypectomy of eligible lesions will be performed in a gas distended colon. Hot and cold resection techniques will be utilized. Submucosal fluid injection with a solution containing hydroxyethyl starch, dilute epinephrine and a contrast agent may be used with conventional techniques for large (≥1cm) and/or flat lesions. There will be no limit to the amount of submucosal injection used.
  Arms: Conventional resection
Procedure: Standard polypectomy — Standard polypectomy will be performed for diminutive (<6mm), pedunculated and semi-pedunculated lesions that do not fall under the inclusion criteria for the study. These lesions will be removed in a gas distended colon with a 9mm firm, thin wire cold snare or snare electrocautery for large (≥1cm) lesions.

SUMMARY:
The aim of this study is to compare the efficacy of underwater resection (polypectomy) versus conventional polypectomy techniques for small and large colorectal lesions identified during colonoscopy.

DETAILED DESCRIPTION:
Conventional endoscopic resection of small and large (≥1cm) colorectal lesions is well established and performed with the colon fully distended with gas. Conventional polypectomy is effective, but the rate of incomplete resection is approximately 10%. Incomplete eradication of precancerous lesions contributes to interval colorectal cancer; therefore, alternative techniques for resection that safely and effectively increase the rate of complete resection are important. Underwater resection (UR) of benign colorectal lesions is a novel technique that utilizes the advantages of water aided endoscopic methods and may decrease the incomplete resection rate of small and large non-pedunculated lesions.

The investigators propose the hypothesis that small (6-9mm) and large (≥1cm) non-pedunculated neoplastic colorectal lesions resected by UR (partially distended, water filled lumen without submucosal fluid injection), will significantly decrease the incomplete resection rate (IRR) compared to conventional polypectomy performed in a gas distended lumen.

Small (6-9mm) and large (≥1cm) non-pedunculated benign neoplastic colorectal lesions identified during screening, surveillance, diagnostic or therapeutic colonoscopy will be randomized to conventional polypectomy (in a gas distended lumen with or without submucosal fluid injection) versus UR (partially distended, water filled lumen without submucosal injection) at the patient level. Small (6-9mm) lesions will be removed with a 9mm firm, thin wire cold snare and large (≥1cm) lesions will be removed by snare electrocautery. Efforts to remove lesions en bloc with a small rim of normal mucosa will be made, although some larger lesions (≥2cm) may require piecemeal resection. Submucosal fluid injection with a solution may be used with conventional techniques for large and/or flat lesions. Post-polypectomy incomplete resection rates will be assessed from 4 quadrant biopsies obtained around the resection site immediately post-resection.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old) male and female patients.
* Scheduled for outpatient colonoscopy.
* Patient able to provide informed consent.
* Benign, small (6-9mm) and large (≥1cm) non-pedunculated colorectal lesions.

Exclusion Criteria:

* Diminutive (≤5mm) and pedunculated polyps.
* Lesions suspected of harboring deep submucosal invasion.
* Patients who decline to participate or are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-09; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Incomplete resection rate (histologic) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Yen, MD, Principal Investigator — VA Northern California Health Care System
Locations (1):
- Sacramento VA Medical Center (VANCHCS), Mather, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pohl H, Srivastava A, Bensen SP, Anderson P, Rothstein RI, Gordon SR, Levy LC, Toor A, Mackenzie TA, Rosch T, Robertson DJ. Incomplete polyp resection during colonoscopy-results of the complete adenoma resection (CARE) study. Gastroenterology. 2013 Jan;144(1):74-80.e1. doi: 10.1053/j.gastro.2012.09.043. Epub 2012 Sep 25. PMID 23022496
- [Background] Binmoeller KF, Weilert F, Shah J, Bhat Y, Kane S. "Underwater" EMR without submucosal injection for large sessile colorectal polyps (with video). Gastrointest Endosc. 2012 May;75(5):1086-91. doi: 10.1016/j.gie.2011.12.022. Epub 2012 Feb 25. PMID 22365184
- [Derived] Yen AW, Leung JW, Wilson MD, Leung FW. Underwater versus conventional endoscopic resection of nondiminutive nonpedunculated colorectal lesions: a prospective randomized controlled trial (with video). Gastrointest Endosc. 2020 Mar;91(3):643-654.e2. doi: 10.1016/j.gie.2019.09.039. Epub 2019 Oct 16. PMID 31628954